CLINICAL TRIAL: NCT07307027
Title: Could a Stepwise Enteral Nutritional Algorithm Affect Patient's Outcome in Pediatric Intensive Care Units? An Interventional Study
Brief Title: Stepwise Enteral Nutritional Algorithm and Patient Outcomes in Pediatric Intensive Care Units
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MD331/2024
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Enteral Nutrition; Enteral Nutrition Feeding; Enteral Nutrition Intolerance in Critically Ill Patients
Keywords: enteral nutrition in critically ill; EN

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental pre-post implementation study. Participants are recruited sequentially in two phases: a baseline "pre-implementation" cohort managed with standard care, followed by a "post-implementation" cohort managed using the new stepwise enteral nutritional algorithm.
Masking Description: This is an open-label study. Participants, care providers, and investigators are aware of the assigned intervention (standard care vs. nutritional algorithm) due to the nature of the feeding protocol implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation phase (Standard Care) (No Intervention): This group consists of 40 patients recruited consecutively before the introduction of the new nutritional algorithm. Patients in this arm receive the standard nutritional care practices currently used in the Pediatric Intensive Care Unit without the standardized stepwise protocol.
- Post-implementation (Intervention) (Experimental): This group consists of 40 patients recruited after the implementation of the standardized stepwise Enteral Nutritional (EN) algorithm. Patients in this arm are managed according to the specific guidelines for feeding initiation, advancement, and intolerance management defined in the study protocol.
  Interventions: Other: Stepwise Enteral Nutritional Algorithm

INTERVENTIONS:
Other: Stepwise Enteral Nutritional Algorithm — A standardized, stepwise protocol for the initiation, advancement, and maintenance of enteral nutrition in critically ill children. It includes specific guidelines for caloric targets, managing feeding intolerance (vomiting, diarrhea, distention), and standardized fasting times for procedures to minimize interruptions.
  Other Names: Standardized nutritional protocol; Enteral nutritional algorithm
  Arms: Post-implementation (Intervention)

SUMMARY:
The aim of the study to evaluate the effectiveness and patient's outcome after implementing enteral nutrition algorithm designed to achieve optimal enteral nutrition delivery in the pediatric intensive care unit and to evaluate the effect of implementing this protocol on critically ill patient's individual's outcome.

DETAILED DESCRIPTION:
The aim of the study to evaluate the effectiveness and patient's outcome after implementing enteral nutrition algorithm designed to achieve optimal enteral nutrition delivery in the pediatric intensive care unit and to evaluate the effect of implementing this protocol on critically ill patient's individual's outcome. Critically ill children in Pediatric Intensive Care Units (PICUs) are particularly vulnerable to malnutrition due to limited body reserves, high metabolic stress, and the catabolic nature of critical illness. While Enteral Nutrition (EN) is the preferred method of nutrient delivery, its optimal implementation is frequently hindered by avoidable barriers and interruptions, such as prolonged fasting for procedures or conservative management of gastrointestinal intolerance. Delays in initiating and advancing EN are associated with failure to reach energy goals and poorer clinical outcomes. This study hypothesizes that implementing a uniform, stepwise nutritional algorithm will decrease avoidable EN interruptions, optimize nutrient delivery, and improve patient outcomes.

Study Design and Methods: This is a prospective, interventional study utilizing a pre/post-implementation design to evaluate the efficacy of a standardized feeding protocol. The study will be conducted at the Pediatric Intensive Care Units of Ain Shams University Children's Hospital.

The study is divided into two distinct phases:

Pre-implementation Phase: Baseline data will be collected on 40 consecutively recruited patients managed under the unit's standard care practices without the specific algorithm.

Post-implementation Phase: A new, stepwise nutritional algorithm will be implemented for a subsequent cohort of 40 patients.

The Intervention (Stepwise Nutritional Algorithm): The intervention involves a structured protocol for nutritional assessment, feeding initiation, advancement, and management of intolerance.

Key components of the algorithm include:

Nutritional Assessment: All patients undergo anthropometric assessment (weight, height/length, MUAC) and screening using the STRONGkids tool and WHO/CDC growth charts upon admission.

Caloric Targets: Energy requirements are calculated using WHO guidelines or the Schofield equation (for sedated/ventilated patients), and protein goals are set based on ASPEN guidelines (ranging from 1.5 to 3 g/kg/day depending on age).

Initiation of Feeding: Enteral feeding is to be initiated within 4 hours of admission absent contraindications (e.g., hemodynamic instability, bowel obstruction).

Feeding Strategy:

Infants <1 year: Expressed breast milk is the preferred first line; if unavailable, standard infant formula is used.

Advancement: Feeding typically starts at 20 ml/kg/day divided every 3 hours. If tolerated, it is advanced by 2 ml/kg/feed every 3 hours until target goals are met.

Management of Intolerance: The protocol provides specific definitions and management steps for intolerance symptoms:

Emesis: Defined as ≥2 episodes/24 hrs. Diarrhea: Defined as >3 episodes of loose stool/24 hrs. Abdominal Distention: Defined as an increase in abdominal girth by >2 cm from baseline for 2 consecutive feds.

Procedural Fasting: The algorithm standardizes fasting times (NPO) prior to procedures to minimize unnecessary interruptions (e.g., 4 hours for elective intubation, 6 hours for surgical procedures under GA).

Data Collection and Comparison: Outcomes will be compared between the pre-implementation and post-implementation cohorts.

Data collection includes:

Nutritional Metrics: Time from admission to EN initiation, time to reach target energy goals, and the frequency and duration of EN interruptions.

Clinical Outcomes: Duration of mechanical ventilation, length of PICU stay, and patient survival/mortality.

Safety: Incidence of feeding intolerance (vomiting, diarrhea, distention) and aspiration risks.

Statistical Analysis: Data will be analyzed using SPSS version 23. Quantitative data will be compared using Student's T-test or Mann-Whitney tests, while qualitative data will be analyzed using Chi-square or Fisher's exact tests. A p-value of ≤0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill infants and children admitted to the Pediatric Intensive Care Units.
* Age range from 1 month to 16 years (specifically males up to 14 years and females up to 16 years).

Exclusion Criteria:

* Patients who are discharged or died within 24 hours of admission.
* Patients with acute pancreatitis.
* Patients with esophageal perforation.
* Patients with a known metabolic disorder.
* Patients requiring a ketogenic diet.
* Patients with Short Bowel Syndrome.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Time to reach target energy goals | From date of admission until energy goals are reached, assessed up to 28 days.
  The duration (measured in days) required for the patient to achieve 100% of their calculated daily caloric target via enteral nutrition. Caloric targets are determined using FAO/WHO/UNU estimated energy requirements or the Schofield equation for sedated/ventilated patients.
Number of enteral nutrition interruptions | From date of admission up to 28 days.
  The total count of episodes where enteral feeding was temporarily or permanently stopped. An interruption is defined as the cessation of feeding for reasons such as hemodynamic instability, medical procedures, or aspiration risk.

SECONDARY OUTCOMES:
Length of Pediatric Intensive Care Unit stay | From date of admission assessed up to 28 days.
  The total duration (in days) a patient remains in the PICU from admission to discharge. This measure is compared between the pre-implementation and post-implementation groups to evaluate if the stepwise nutritional algorithm reduces the length of stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share